CLINICAL TRIAL: NCT04245059
Title: Safety Study Based on Transcranial Electrical Stimulation in Chile: a Case Series Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Corporación de Rehabilitación Club de Leones Cruz del Sur (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CorporacionRCLCS0002
Record Dates: First submitted 2020-01-22; First posted 2020-01-28 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Healthy Subjects
Keywords: transcranial electrical stimulation; transcranial direct current stimulation; motor cortex; motor performance; secondary effects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcranial Direct Current Stimulation (Experimental): Each subject will receive transcranial electrical stimulation at primary motor cortex in both hemispheres. The pilot program will include 12 sessions with a frequency of 3 times per week during 4 weeks. Therefore, during tDCS sessions, subjects will receive stimulation for 20 minutes with a current of 2.0 milliamp using 6x4 cm electrodes. The participants will also complete a set of manual dexterity, grip and pinch tests bilaterally at baseline and post-intervention to determine if the subject responds to tDCS. Thus, each session will be monitored on safety aspects of the subjects with emphasis on skin disorders and other possible side effects of tDCS.
  Interventions: Device: Multi-channel Transcranial direct current stimulation

INTERVENTIONS:
Device: Multi-channel Transcranial direct current stimulation — A commercial tDCS device will be use in this study. The device is a wireless multi-channel transcranial direct current stimulator that incorporates an 8-channel headcap for stimulation through gel electrodes or classic sponge electrodes. The device is integrated with a user interface for the configuration and monitoring of the stimulus parameters and a fast multifocal simulation of the tDCS electric field using an advanced brain model

SUMMARY:
Transcranial direct current stimulation (tDCS) is a non-invasive neuromodulation technique that delivers low-intensity, direct current to cortical areas facilitating or inhibiting spontaneous neuronal activity. It has been used to improve cognitive functions such as memory, language, and attention. Research has also shown that tDCS on motor cortex can improve motor performance.

TDCS secondary effects have been measured in several studies. The most frequent secondary effects described in literature are a mild tingling sensation, moderate fatigue, itching sensation, slight burning and mild pain sensation under the electrodes during the stimulation.

The present study is focused in evaluate the safety of a transcranial direct current stimulation (TDCS) service by measuring secondary effects incidence in a group of healthy subjects. In addition, manual dexterity and upper limb strength will be measure to identify improvement in motor performance after intervention.

DETAILED DESCRIPTION:
Transcranial electrical stimulation (tES) is a neurophysiological technique capable of modulating the excitability of the neuronal tissue of the central and peripheral nervous system through the application, for a finite time length, of an electrical field. This electric field is generated by the application of weak electrical currents through the scalp and into the brain. It has been demonstrated in recent years that the technique is safe and beneficial if used within the known bounds of intensity, density and duration.

The tES technique is classified into three types according to the waveform of the stimulation current that is applied: Transcranial direct current stimulation (tDCS),Transcranial Alternating Current Stimulation (tACS) and Transcranial random noise stimulation (tRNS). Additionally, the Sham mode can be used for controlled experiments.

TDCS is a neuromodulatory technique that delivers low-intensity, direct current to cortical areas facilitating or inhibiting spontaneous neuronal activity. In general, the current is injected into the brain (anodal stimulation) over a cortical region leading to excitatory effects; and collected from the brain (cathodal stimulation) leading to inhibitory effects. tDCS produces short term effects on neuronal excitability, and long lasting plastic after/effects involving synaptic modification.

Research has shown that applying anodal tDCS to the non-dominant motor cortex can improve motor performance for the non-dominant hand, presumably by means of changes in synaptic plasticity between neurons. Other studies suggest improvement on cognitive functions such as memory, language, and attention after a tDCS program.

TDCS secondary effects have been measured in several studies. The most frequent secondary effects described in literature are a mild tingling sensation, moderate fatigue, itching sensation, slight burning and mild pain sensation under the electrodes during the stimulation. A visual sensation, associated with switching on and off the stimulation, have been also described. Less frequent are the difficulties in concentrating, headache, felt nervous or overexcited and nausea after the stimulation.

The present study is focused in evaluate the safety of a TDCS pilot program by measuring secondary effects incidence in a group of healthy subjects. In addition, manual dexterity and upper limb strength will be measure to identify improvement in motor performance after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Both gender
* Informed consent accepted
* Adults

Exclusion Criteria:

* Neurological diseases
* Mental diseases
* Injuries in the scalp skin
* Inflammatory tegumentary diseases
* Migraines
* Medication or substances affecting central nervous system
* Presence of chronic diseases
* Presence of degenerative diseases
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of block and box test score | Baseline, 4 weeks
  Change of the Box and Block test score, it's a measure of the number of blocks the subject can move in 1 minute, between the beginning (T0) and immediately after the end of treatment (T1). Range of score 0-120. A positive change represents improved performance on Box and Blocks test.
Change of Side effect checklist for transcranial direct current stimulation | Baseline, 4 weeks
  A checklist that records side effect after TDCS sessions including fatigue, headache or dizziness, nausea, and a itching sensation in the stimulation area.

SECONDARY OUTCOMES:
Change of nine hole peg test score | Baseline, 4 weeks
  The Nine Hole Pegs technique is a simple manual dexterity test, commonly used in ergotherapy. The participant tries to place 9 pegs in a 9 holes perforated plate, and then tries to remove them as quickly as possible. The hand must stay in a depression within the plate, thereby insuring a constant distance between the hand and the pegs.
Change of grip strength measurement | Baseline, 4 weeks
  Change of value of kilogram - force (kgf) measured with a handheld dynamometer on a single grip test of maximum contraction for 3 seconds.
Change of pinch strength measurement | Baseline, 4 weeks
  Change of value of kilogram - force (kgf) measured with a handheld dynamometer on a single pinch test of maximum contraction for 3 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Patricio E Barría Aburto, MSc., Principal Investigator — Corporación de Rehabilitacion Club de Leones Cruz del Sur; Karim S Baleta Abarza, Lic., Principal Investigator — Corporación de Rehabilitacion Club de Leones Cruz del Sur
Locations (1):
- Corporación de Rehabilitación Club de Leones Cruz del Sur, Punta Arenas, Region of Magallanes, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brunoni AR, Nitsche MA, Bolognini N, Bikson M, Wagner T, Merabet L, Edwards DJ, Valero-Cabre A, Rotenberg A, Pascual-Leone A, Ferrucci R, Priori A, Boggio PS, Fregni F. Clinical research with transcranial direct current stimulation (tDCS): challenges and future directions. Brain Stimul. 2012 Jul;5(3):175-195. doi: 10.1016/j.brs.2011.03.002. Epub 2011 Apr 1. PMID 22037126
- [Background] Vines BW, Cerruti C, Schlaug G. Dual-hemisphere tDCS facilitates greater improvements for healthy subjects' non-dominant hand compared to uni-hemisphere stimulation. BMC Neurosci. 2008 Oct 28;9:103. doi: 10.1186/1471-2202-9-103. PMID 18957075
- [Background] Almousa A, Alajaji R, Alaboudi M, Al-Sultan F, Bashir S. Safety of Transcranial Direct Current Stimulation of Frontal, Parietal, and Cerebellar Regions in Fasting Healthy Adults. Behav Sci (Basel). 2018 Sep 10;8(9):81. doi: 10.3390/bs8090081. PMID 30201910
- [Background] Paulus W. Transcranial electrical stimulation (tES - tDCS; tRNS, tACS) methods. Neuropsychol Rehabil. 2011 Oct;21(5):602-17. doi: 10.1080/09602011.2011.557292. Epub 2011 Aug 5. PMID 21819181